CLINICAL TRIAL: NCT06936956
Title: The Effect of Acupressure on Polyneuropathy-related Pain and Sleep Quality in Patients With Type 2 Diabetes
Brief Title: The Effect of Acupressure on Polyneuropathy-related Pain and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Fatma Gündüz Oruç, Dr. Öğr. Üyesi, Giresun University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GRU-SBF-FGO-01
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes
Keywords: Acupressure, diabetes, nursing, polyneuropathy, sleep quality
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Polyneuropathies; Sleep Initiation and Maintenance Disorders | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure group (Experimental): Particiants in this group received acupressure application.
  Interventions: Other: Acupressure
- Control group (No Intervention): Participants in this group did not receive any intervention.

INTERVENTIONS:
Other: Acupressure — Acupressure is a noninvasive type of acupuncture. It is applied using fingers, joints or a suitable acupressure tool.
  Arms: Acupressure group

SUMMARY:
This study aimed to determine the effect of acupressure on polyneuropathy-related pain and sleep quality in patients with type 2 diabetes. A randomized controlled experimental design was employed in the study. The study sample consisted of 86 patients with type 2 diabetes (44 in the acupressure group and 42 in the control group) who met the inclusion criteria and agreed to participate. Participants were randomly assigned to either the experimental or control group. The experimental group received six sessions of acupressure over six consecutive days, while the control group received no intervention. Data were collected using a personal information form, the Pain Quality Assessment Scale (PQAS), and the Pittsburgh Sleep Quality Index (PSQI). Statistical analyses were conducted using SPSS for Windows 22. Acupressure was found to reduce polyneuropathy-related pain and enhance sleep quality in patients with type 2 diabetes. Therefore, acupressure may be considered an alternative nursing intervention for individuals with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Were between the ages of 18-65 years old
* Resided in the city center
* Had no additional diseases that could cause sensory neuropathy, such as peripheral arterial disease, peripheric vein disease, nervous system diseases, benign or malign tumor, chemotherapy history, carpal tunnel syndrome, and arthritis.
* Had no clotting or bleeding disorders
* Were not undergoing dialysis treatment during the study period
* Had no ulcers, physical deformities or foot calluses
* Had no history of analgesic medication, except for medication used for DPN
* Had no physical diseases, cognitive deficiencies or psychiatric disease diagnosis that would prevent understanding of the questions on the scales used for data collection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Pain Quality Assessment Scale (PQAS) | 6 days
  This scale was originally developed by Galer et al. as the Neuropathic Pain Scale and its validity was confirmed with multiple sclerosis patients (Galer&Jensen 1997). However, this original scale does not include allodynia and paroxysmal pain characteristics, which are common in neuropathic pain syndromes. Jensen et al. developed the Pain Quality Assessment Scale (PQAS) by adding 10 items related to the quality of neuropathic pain, and its validity was confirmed by measuring the neuropathic pain due to carpal tunnel syndrome (Cronbach's alpha 0.87-0.98) (Jense et al.,2006). Şahin et al. adapted the final version of the scale for Turkish society and reported that it is reliable to be used for the cases of diseases with neuropathic pain (Şahin et al., 2010). For the PQAS, it is recommended that no total score be calculated; rather, the three subscales are scored from 0 to 10. In this study, the Cronbach's alpha values were 0.836 for the paroxysmal pain subscale, 0.624 for the surface pa
Pittsburgh Quality of Sleep Index (PQSI) | 6 days
  This questionnaire was developed by Buysse et al. and was confirmed to have a high internal consistency (Cronbach's alpha=0.75), test-retest reliability, and validity (Buyyse et al., 1989). A study was conducted to confirm the Turkish validity and reliability of the questionnaire (Cronbach alpha=0.660) (Ağargün&Anlar 1996). Each item of the questionnaire is scored between 0 and 3, and the total PQSI score, which ranges between 0 and 21, is obtained by adding the subscale scores. A PSQI score between 0 and 4 indicates a good quality of sleep, while a score between 5 and 21 indicates a bad quality of sleep (Ağargün&Anlar 1996). In the present study, Cronbach's alpha value was 0.576 for the total PSQI.

CONTACTS AND LOCATIONS:
Overall Officials: Elanur YILMAZ KARABULUTLU Professör, pHD, Study Director — Erzurum Technical University
Locations (1):
- Endocrinology Clinic and Outpatient Clinic of a Atatürk University Hospital, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not want my data to be used by other researchers